CLINICAL TRIAL: NCT02694523
Title: BI 655066/ABBV-066 (Risankizumab) Versus Adalimumab in a Randomized, Double Blind, Parallel Group Trial in Moderate to Severe Plaque Psoriasis to Assess Safety and Efficacy After 16 Weeks of Treatment and After Inadequate Adalimumab Treatment Response (IMMvent)
Brief Title: BI 655066/ABBV-066 (Risankizumab) Compared to Active Comparator (Adalimumab) in Patients With Moderate to Severe Chronic Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M16-010; 2015-003623-65 (EudraCT Number); 1311.30 (Other: Boehringer Ingelheim)
Record Dates: First submitted 2016-02-24; First posted 2016-02-29 (Estimated); Results first posted 2019-05-28 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Psoriasis
Keywords: Psoriasis; Skin Diseases; Skin Diseases, Papulosquamous; Adalimumab; Anti-Inflammatory Agents; ABBV-066; BI 655066; Risankizumab
MeSH Terms: conditions — Psoriasis; Skin Diseases; Skin Diseases, Papulosquamous | interventions — risankizumab; Adalimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adalimumab (Part A) (Active Comparator): Participants randomized to receive double-blind (DB) adalimumab 80 mg by subcutaneous (SC) injection at Week 0, then 40 mg at Week 1 and every 2 weeks for 15 weeks (Part A).
  Interventions: Biological: adalimumab; Drug: placebo for risankizumab
- Risankizumab (Part A) (Experimental): Participants randomized to receive risankizumab at Weeks 0 and 4 (Part A).
  Interventions: Drug: risankizumab; Biological: placebo for adalimumab

INTERVENTIONS:
Drug: risankizumab — Risankizumab administered by subcutaneous (SC) injection
  Other Names: BI 655066; ABBV-066; SKYRIZI
  Arms: Risankizumab (Part A)
Biological: adalimumab — Adalimumab pre-filled syringe, administered by subcutaneous (SC) injection
  Other Names: Humira; ABT-D2E7
  Arms: Adalimumab (Part A)
Drug: placebo for risankizumab — Placebo risankizumab administered by subcutaneous (SC) injection
  Arms: Adalimumab (Part A)
Biological: placebo for adalimumab — Placebo for adalimumab pre-filled syringe, administered by subcutaneous (SC) injection
  Arms: Risankizumab (Part A)

SUMMARY:
This is a randomized double blind, double dummy, active comparator controlled, parallel design study that is performed to assess the safety and efficacy of BI 655066/ABBV-066 (risankizumab) compared to adalimumab to support registration for the treatment of moderate to severe chronic plaque psoriasis in adult patients.

DETAILED DESCRIPTION:
This study consists of 2 parts (Part A and Part B).

Part A:

* Participants were randomized to receive either risankizumab or adalimumab.

Part B:

* Participants who received risankizumab in Part A continued to receive risankizumab in Part B
* Adalimumab nonresponders (<PASI 50 at Week 16) switched to risankizumab in Part B;
* Adalimumab responders (PASI 90 at Week 16) continued to received adalimumab in Part B;
* Adalimumab inadequate responders (PASI 50 to <PASI 90) were rerandomized to receive either risankizumab or adalimumab in Part B.

ELIGIBILITY:
Inclusion criteria:

* Male or female patients. Women of childbearing potential* must be ready and able to use highly effective methods of birth control per ICH M3(R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. A list of contraception methods meeting these criteria is provided in the patient information.

  *Women of childbearing potential are defined as:
  * having experienced menarche and
  * not postmenopausal (12 months with no menses without an alternative medical cause) and
  * not permanently sterilized (e.g., tubal occlusion, hysterectomy, bilateral oophorectomy or bilateral salpingectomy).
* Age ≥ 18 years at screening
* Have a diagnosis of chronic plaque psoriasis (with or without psoriatic arthritis) for at least 6 months before the first administration of study drug. Duration of diagnosis may be reported by the patient.
* Have stable moderate to severe chronic plaque psoriasis with or without psoriatic arthritis at both Screening and Baseline (Randomization):

  * Have an involved body surface area (BSA) ≥ 10% and
  * Have a Psoriasis Area and Severity Index (PASI) score ≥ 12 and
  * Have a static Physician Global Assessment (sPGA) score of ≥ 3.
* Must be candidates for systemic therapy or phototherapy for psoriasis treatment, as assessed by the investigator
* Must be candidates for treatment with adalimumab (Humira®) according to local label as confirmed by the investigator.
* Signed and dated written informed consent prior to admission to the study in accordance with GCP and local legislation

Exclusion criteria:

* Patients with

  * non-plaque forms of psoriasis (including guttate, erythrodermic, or pustular)
  * current drug-induced psoriasis (including an exacerbation of psoriasis from beta blockers, calcium channel blockers, or lithium)
  * active ongoing inflammatory diseases other than psoriasis that might confound trial evaluations according to investigator's judgment
* Previous exposure to ABBV-066
* Previous exposure to adalimumab (Humira®)
* Currently enrolled in another investigational study or less than 30 days or more from screening since completing another investigational drug or device study.
* Use of any restricted medication or any drug considered likely to interfere with the safe conduct of the study.
* Major surgery performed within 12 weeks prior to randomization or planned within 12 months after screening (e.g. hip replacement, removal aneurysm, stomach ligation).
* Known chronic or relevant acute infections, such as active tuberculosis (TB), human immunodeficiency virus (HIV) or viral hepatitis; QuantiFERON® TB test or purified protein derivative (PPD) skin test will be performed according to local labelling for Humira®. If the result is positive, patients may participate in the study if further work up (according to local practice/guidelines) establishes conclusively that the patient has no evidence of active TB. If presence of latent TB is established, then treatment should have been initiated and maintained according to local country guidelines.
* Any documented active or suspected malignancy or history of malignancy within 5 years prior to screening, except appropriately treated basal cell or squamous cell carcinoma of the skin or in situ carcinoma of uterine cervix.
* Evidence of a current or previous disease, medical condition (including chronic alcohol or drug abuse) other than psoriasis, surgical procedure (i.e., organ transplant), medical examination finding (including vital signs and electrocardiogram [ECG]), or laboratory value at the Screening Visit outside the reference range that in the opinion of the investigator is clinically significant and would make the study participant unreliable to adhere to the protocol or to complete the trial, compromise the safety of the patient, or compromise the quality of the data.
* History of allergy/hypersensitivity to a systemically administered biologic agent or its excipients
* Women who are pregnant, nursing, or who plan to become pregnant while in the trial
* Previous enrolment in this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 684 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim

REFERENCES:
- [Background] Reich K, Gooderham M, Thaci D, Crowley JJ, Ryan C, Krueger JG, Tsai TF, Flack M, Gu Y, Williams DA, Thompson EHZ, Paul C. Risankizumab compared with adalimumab in patients with moderate-to-severe plaque psoriasis (IMMvent): a randomised, double-blind, active-comparator-controlled phase 3 trial. Lancet. 2019 Aug 17;394(10198):576-586. doi: 10.1016/S0140-6736(19)30952-3. Epub 2019 Jul 4. PMID 31280967
- [Derived] Hsieh CY, Hsu FL, Tsai TF. Comparison of Drug-Free Remission after the End of Phase III Trials of Three Different Anti-IL-23 Inhibitors in Psoriasis. Dermatol Ther (Heidelb). 2024 Sep;14(9):2607-2620. doi: 10.1007/s13555-024-01229-6. Epub 2024 Jul 29. PMID 39073712
- [Derived] Lebwohl MG, Soliman AM, Yang H, Wang J, Hagan K, Padilla B, Pinter A. Impact of Risankizumab on PASI90 and DLQI0/1 Duration in Moderate-to-Severe Psoriasis: A Post Hoc Analysis of Four Phase 3 Clinical Trials. Dermatol Ther (Heidelb). 2022 Feb;12(2):407-418. doi: 10.1007/s13555-021-00660-3. Epub 2021 Dec 18. PMID 34921669
- [Derived] Suleiman AA, Khatri A, Oberoi RK, Othman AA. Exposure-Response Relationships for the Efficacy and Safety of Risankizumab in Japanese Subjects with Psoriasis. Clin Pharmacokinet. 2020 May;59(5):575-589. doi: 10.1007/s40262-019-00829-2. PMID 31667790
- [Derived] Suleiman AA, Minocha M, Khatri A, Pang Y, Othman AA. Population Pharmacokinetics of Risankizumab in Healthy Volunteers and Subjects with Moderate to Severe Plaque Psoriasis: Integrated Analyses of Phase I-III Clinical Trials. Clin Pharmacokinet. 2019 Oct;58(10):1309-1321. doi: 10.1007/s40262-019-00759-z. PMID 31054118
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 684 subjects were enrolled; 79 subjects failed screening and are excluded from the analyses.
Groups:
- Risankizumab (Part A): Participants randomized to receive double-blind (DB) risankizumab 150 mg by subcutaneous (SC) injection at Weeks 0 and 4 (Part A).
- Risankizumab/Risankizumab (Part B): Participants randomized to receive double-blind (DB) risankizumab in Part A continued to receive risankizumab 150 mg by subcutaneous (SC) injection at Weeks 16, and 28 (Part B).
- Adalimumab/Adalimumab (Part B): Participants who were responders after receiving adalimumab in Part A continued to receive adalimumab 40 mg by subcutaneous (SC) injection every other week through Week 41 (Part B).
- Adalimumab/Risankizumab (Part B): Participants who were nonresponders after receiving adalimumab in Part A switched to risankizumab 150 mg by subcutaneous (SC) injection at Weeks 16, 20, and 32 (Part B).
- Adalimumab/Rerandomized to Adalimumab (Part B): Participants who were inadequate responders after receiving adalimumab in Part A and rerandomized to continue to receive adalimumab 40 mg by subcutaneous (SC) injection every 2 weeks through Week 41 (Part B).
- Adalimumab/Rerandomized to Risankizumab (Part B): Participants who were inadequate responders after receiving adalimumab in Part A and rerandomized to receive risankizumab 150 mg by subcutaneous (SC) injection at Weeks 16, 20, and 32 (Part B).
Period: Part A
Arm/Group | Adalimumab (Part A) | Risankizumab (Part A) | Risankizumab/Risankizumab (Part B) | Adalimumab/Adalimumab (Part B) | Adalimumab/Risankizumab (Part B) | Adalimumab/Rerandomized to Adalimumab (Part B) | Adalimumab/Rerandomized to Risankizumab (Part B)
Started | 304 | 301 | 0 | 0 | 0 | 0 | 0
Completed | 291 | 294 | 0 | 0 | 0 | 0 | 0
Not Completed | 13 | 7 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 7 | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 1 | 1 | 0 | 0 | 0 | 0 | 0
Period: Part B
Arm/Group | Adalimumab (Part A) | Risankizumab (Part A) | Risankizumab/Risankizumab (Part B) | Adalimumab/Adalimumab (Part B) | Adalimumab/Risankizumab (Part B) | Adalimumab/Rerandomized to Adalimumab (Part B) | Adalimumab/Rerandomized to Risankizumab (Part B)
Started | 0 | 0 | 294 (Participants who received risankizumab in Part A continued to received risankizumab in Part B) | 144 (Adalimumab responders in Part A continued to received adalimumab in Part B) | 38 (Adalimumab nonresponders in Part A switched to risankizumab in Part B) | 56 (Adalimumab inadequate responders in Part A, rerandomized to adalimumab in Part B) | 53 (Adalimumab inadequate responders in Part A, rerandomized to risankizumab in Part B)
Completed | 0 | 0 | 274 | 140 | 34 | 51 | 51
Not Completed | 0 | 0 | 20 | 4 | 4 | 5 | 2
Not completed — Adverse Event | 0 | 0 | 7 | 1 | 1 | 2 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 2 | 3 | 2 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 9 | 0 | 1 | 3 | 0
Not completed — Other | 0 | 0 | 1 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population in Part A (ITT_A): All subjects randomized at Baseline.
Groups:
- Adalimumab (Part A): Participants randomized to receive double blind (DB) adalimumab 80 mg by subcutaneous (SC) injection at Weeks 0, 1, and every other week for 15 weeks (Part A).
- Risankizumab (Part A): Participants randomized to receive double-blind (DB) risankizumab 150 mg by subcutaneous (SC) injection at Weeks 0, 4 (Part A).
- Total: Total of all reporting groups
Arm/Group | Adalimumab (Part A) | Risankizumab (Part A) | Total
Number analyzed (Participants) | 304 | 301 | 605
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.0 (13.09) | 45.3 (13.79) | 46.2 (13.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 91 | 183
  Male | 212 | 210 | 422
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 59 | 44 | 103
  Not Hispanic or Latino | 245 | 257 | 502
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 35 | 41 | 76
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 11 | 17
  White | 263 | 245 | 508
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving 90% Improvement in Psoriasis Area and Severity Index (PASI) Score (PASI90) at Week 16 (Part A)
Description: PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign was assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI90 is defined as at least a 90% reduction in PASI score compared with the Baseline PASI score. The percent reduction in score is calculated as (PASI score at Baseline - score at follow-up visit) / PASI score at Baseline * 100. Nonresponder imputation (NRI) was used for missing data.
Time Frame: Week 16
Population: Intent-to-treat population in Part A (ITT_A): All subjects randomized at Baseline.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab (Part A) | Risankizumab (Part A)
Number analyzed (Participants) | 304 | 301
percentage of participants | 47.4 | 72.4
Statistical Analysis 1: Comparison: Adalimumab (Part A) vs Risankizumab (Part A); P-value calculated according to the Cochran-Mantel-Haenszel test adjusted for baseline weight (≤100 kg vs >100 kg) and prior exposure to tumor necrosis factor (TNF) antagonists (0 vs ≥1); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; difference in percentage of participants = 24.9, 95% CI 2-sided [17.5 to 32.4]

2. Primary Outcome: Percentage of Participants Achieving Static Physician Global Assessment (sPGA) Score of Clear or Almost Clear at Week 16 (Part A)
Description: The sPGA is an assessment by the investigator of the overall disease severity at the time of evaluation. Erythema (E), induration (I), and desquamation (D) are scored on a 5-point scale ranging from 0 (none) to 4 (severe). The sPGA ranges from 0 to 4, and is calculated as Clear (0) = 0 for all three; Almost clear (1) = mean >0, <1.5; Mild (2) = mean ≥1.5, <2.5; Moderate (3) = mean ≥2.5, <3.5; and Severe (4) = mean ≥3.5. NRI was used for missing data.
Time Frame: Week 16
Population: ITT_A population.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab (Part A) | Risankizumab (Part A)
Number analyzed (Participants) | 304 | 301
percentage of participants | 60.2 | 83.7
Statistical Analysis 1: Comparison: Adalimumab (Part A) vs Risankizumab (Part A); P-value calculated according to the Cochran-Mantel-Haenszel test adjusted for baseline weight (≤100 kg vs >100 kg) and prior exposure to TNF antagonists (0 vs ≥1); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; difference in percentage of participants = 23.3, 95% CI 2-sided [16.6 to 30.1]

3. Primary Outcome: Percentage of Participants Who Were Re-Randomized to Receive Either Adalimumab or Risankizumab in Part B Achieving PASI90 at Week 44 (Part B)
Description: PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign was assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI90 is defined as at least a 90% reduction in PASI score compared with the Baseline PASI score. The percent reduction in score is calculated as (PASI score at Baseline - score at follow-up visit) / PASI score at Baseline * 100. NRI was used for missing data.
Time Frame: Week 44
Population: Intent-to-treat population in Part B who were re-randomized (ITT_B_RR): All subjects who started with adalimumab at Baseline and were re-randomized at Week 16
Measure: Number; unit: percentage of participants
Groups:
- Adalimumab/Rerandomized to Adalimumab (Part B): Participants who were inadequate responders after receiving adalimumab in Part A, and rerandomized to continue to receive adalimumab 40 mg by subcutaneous (SC) injection every 2 weeks through Week 41 (Part B).
- Adalimumab/Rerandomized to Risankizumab (Part B): Participants who were inadequate responders after receiving adalimumab in Part A, and rerandomized to receive risankizumab 150 mg by subcutaneous (SC) injection at Weeks 16, 20, and 32 (Part B).
Arm/Group | Adalimumab/Rerandomized to Adalimumab (Part B) | Adalimumab/Rerandomized to Risankizumab (Part B)
Number analyzed (Participants) | 56 | 53
percentage of participants | 21.4 | 66.0
Statistical Analysis 1: Comparison: Adalimumab/Rerandomized to Adalimumab (Part B) vs Adalimumab/Rerandomized to Risankizumab (Part B); [analysis description as in outcome 2, analysis 1]; Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; difference in percentage of participants = 45.0, 95% CI 2-sided [28.9 to 61.1]

4. Secondary Outcome: Percentage of Participants Achieving PASI75 at Week 16 (Part A)
Description: PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign was assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI75 is defined as at least a 75% reduction in PASI score compared with the Baseline PASI score. The percent reduction in score is calculated as (PASI score at Baseline - score at follow-up visit) / PASI score at Baseline * 100. NRI was used for missing data.
Time Frame: Week 16
Population: ITT_A population
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab (Part A) | Risankizumab (Part A)
Number analyzed (Participants) | 304 | 301
percentage of participants | 71.7 | 90.7
Statistical Analysis 1: Comparison: Adalimumab (Part A) vs Risankizumab (Part A); [analysis description as in outcome 2, analysis 1]; Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; difference in percentage of participants = 18.9, 95% CI 2-sided [13.0 to 24.9]

5. Secondary Outcome: Percentage of Participants Achieving PASI100 at Week 16 (Part A)
Description: PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign was assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI100 is defined as a 100% reduction in PASI score compared with the Baseline PASI score. The percent reduction in score is calculated as (PASI score at Baseline - score at follow-up visit) / PASI score at Baseline * 100. NRI was used for missing data.
Time Frame: Week 16
Population: ITT_A population
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab (Part A) | Risankizumab (Part A)
Number analyzed (Participants) | 304 | 301
percentage of participants | 23.0 | 39.9
Statistical Analysis 1: Comparison: Adalimumab (Part A) vs Risankizumab (Part A); [analysis description as in outcome 2, analysis 1]; Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; difference in percentage of participants = 16.7, 95% CI 2-sided [9.5 to 23.9]

6. Secondary Outcome: Percentage of Participants Who Were Rerandomized to Receive Either Adalimumab or Risankizumab in Part B Achieving PASI100 at Week 44 (Part B)
Description: as for outcome 5
Time Frame: Week 44
Population: ITT_B_RR population
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab/Rerandomized to Adalimumab (Part B) | Adalimumab/Rerandomized to Risankizumab (Part B)
Number analyzed (Participants) | 56 | 53
percentage of participants | 7.1 | 39.6
Statistical Analysis 1: Comparison: Adalimumab/Rerandomized to Adalimumab (Part B) vs Adalimumab/Rerandomized to Risankizumab (Part B); [analysis description as in outcome 2, analysis 1]; Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; difference in percentage of participants = 32.8, 95% CI 2-sided [18.8 to 46.9]

7. Secondary Outcome: Percentage of Participants Who Were ReRandomized to Receive Either Adalimumab or Risankizumab in Part B Achieving sPGA Score of Clear at Week 44 (Part B)
Description: as for outcome 2
Time Frame: Week 44
Population: ITT_B_RR population
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab/Rerandomized to Adalimumab (Part B) | Adalimumab/Rerandomized to Risankizumab (Part B)
Number analyzed (Participants) | 56 | 53
percentage of participants | 7.1 | 39.6
Statistical Analysis 1: Comparison: Adalimumab/Rerandomized to Adalimumab (Part B) vs Adalimumab/Rerandomized to Risankizumab (Part B); [analysis description as in outcome 2, analysis 1]; Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; difference in percentage of participants = 32.8, 95% CI 2-sided [18.8 to 46.9]

8. Other Pre Specified Outcome: Percentage of Participants Who Were Rerandomized to Receive Either Adalimumab or Risankizumab in Part B Achieving sPGA Score of Clear or Almost Clear at Week 44 (Part B)
Description: as for outcome 2
Time Frame: Week 44
Population: ITT_B_RR population
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab/Rerandomized to Adalimumab (Part B) | Adalimumab/Rerandomized to Risankizumab (Part B)
Number analyzed (Participants) | 56 | 53
percentage of participants | 33.9 | 73.6
Statistical Analysis 1: Comparison: Adalimumab/Rerandomized to Adalimumab (Part B) vs Adalimumab/Rerandomized to Risankizumab (Part B); [analysis description as in outcome 2, analysis 1]; Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; difference in percentage of participants = 38.9, 95% CI 2-sided [22.0 to 55.8]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from first dose of study drug until 15 weeks after the last dose of study drug (up to 48 weeks).
Description: AEs in Part A are defined as events from the first dose of study drug in Part A until prior to the first dose in Part B (Week 16) or up to 15 weeks after the last dose of study drug if the participant discontinued in Part A; AEs in Part B are defined as events from the first dose of study drug in Part B (Week 16) until up to 15 weeks after the last dose of study drug.
Groups:
- Adalimumab/Rerandomized to Adalimumab (Part B): Participants who were inadequate responders after receiving adalimumab in Part A and re-randomized to continue to receive adalimumab 40 mg by subcutaneous (SC) injection every 2 weeks through Week 41 (Part B).
- Adalimumab/Rerandomized to Risankizumab (Part B): Participants who were inadequate responders after receiving adalimumab in Part A and re-randomized to receive risankizumab 150 mg by subcutaneous (SC) injection at Weeks 16, 20, and 32 (Part B).
Arm/Group | Adalimumab (Part A) | Risankizumab (Part A) | Risankizumab/Risankizumab (Part B) | Adalimumab/Risankizumab (Part B) | Adalimumab/Rerandomized to Adalimumab (Part B) | Adalimumab/Rerandomized to Risankizumab (Part B)
All-Cause Mortality (participants affected / at risk) | 2/304 | 1/301 | 0/294 | 0/38 | 0/56 | 0/53
Serious Adverse Events (participants affected / at risk) | 9/304 | 10/301 | 12/294 | 4/38 | 2/56 | 3/53
Other Adverse Events (participants affected / at risk) | 71/304 | 76/301 | 95/294 | 16/38 | 21/56 | 24/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adalimumab (Part A) (N=304) | Risankizumab (Part A) (N=301) | Risankizumab/Risankizumab (Part B) (N=294) | Adalimumab/Risankizumab (Part B) (N=38) | Adalimumab/Rerandomized to Adalimumab (Part B) (N=56) | Adalimumab/Rerandomized to Risankizumab (Part B) (N=53)
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Macrocornea (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Macular hole (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Perirectal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory fume inhalation disorder (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anticoagulation drug level above therapeutic (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abortion induced (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adalimumab (Part A) (N=304) | Risankizumab (Part A) (N=301) | Risankizumab/Risankizumab (Part B) (N=294) | Adalimumab/Risankizumab (Part B) (N=38) | Adalimumab/Rerandomized to Adalimumab (Part B) (N=56) | Adalimumab/Rerandomized to Risankizumab (Part B) (N=53)
Bronchitis (Infections and infestations) | 3 (3) | 4 (4) | 7 (8) | 2 (2) | 3 (3) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 12 (15) | 21 (26) | 34 (44) | 3 (5) | 5 (5) | 4 (6)
Viral upper respiratory tract infection (Infections and infestations) | 24 (29) | 26 (31) | 39 (48) | 9 (14) | 7 (8) | 14 (19)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (12) | 11 (12) | 4 (4) | 0 (0) | 3 (5) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 9 (9) | 6 (6) | 0 (0) | 3 (3) | 2 (3)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 20 (29) | 12 (13) | 6 (7) | 2 (2) | 3 (4) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (6) | 3 (4) | 2 (2) | 1 (1) | 2 (2)
Hypertension (Vascular disorders) | 8 (12) | 1 (1) | 9 (9) | 3 (3) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2016-10-17): https://cdn.clinicaltrials.gov/large-docs/23/NCT02694523/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-12): https://cdn.clinicaltrials.gov/large-docs/23/NCT02694523/SAP_001.pdf